CLINICAL TRIAL: NCT04237077
Title: Impact of a Telephone Coaching Program on Evolution of Autonomy in Subjects Aged 75 Years or More Living at Home
Acronym: Frailcoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PO19126*
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Subjects Aged 75 Years or More Living at Home

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "with telephone coaching program ". (Experimental): subjects aged 75 years or more living at home, with telephone coaching program
  Interventions: Other: telephone coaching program
- Group "without telephone coaching program". (Active Comparator): subjects aged 75 years or more living at home, without telephone coaching program
  Interventions: Other: no telephone coaching program

INTERVENTIONS:
Other: telephone coaching program — telephone coaching program : 7 phone calls by nurse
  Arms: Group "with telephone coaching program ".
Other: no telephone coaching program — no telephone coaching program : 7 phone calls by nurse
  Arms: Group "without telephone coaching program".

SUMMARY:
Since the last few decades, developed societies have been evolving towards a global aging of their populations. This evolution has been accompanied by the problematic of the dependence of aging populations. Dependence is today a challenge posed to social, healthcare or medico-social organizations.

Many studies have shown the positive effect of changes in health (physical activity, nutrition, socialization) on functional abilities of aged subjects. Intervention at subject's home is an easy and inexpensive way to delay the onset of dependence in the elderly population. Health coaching is defined as "a regular series of phone calls between the patient and the health care professional to support and encourage the patient and promote healthy behaviors such as treatment control, healthy eating and physical activity ".

DETAILED DESCRIPTION:
The aim of the study will be evaluate impact of a telephone coaching program on evolution of autonomy in subjects aged 75 years or more living at home

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 75 years or more
* subjects living at home
* subjects able to use phone
* subjects agree to participate to the study

Exclusion Criteria:

* subjects do not speak French

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Autonomy evolution | 12 months
  Evolution of autonomy score between inclusion and 12 months follow up. The autonomy score (on 14 points) is the sum of the Katz's Activities of Daily Living (on 6 points) and the Lawton's Instrumental Activities of Daily Living (on 8 points).
  Katz's Activities of Daily Living comprises 6 items (bathing, dressing, transferring, using the toilet, eating, continence).
  Lawton's Instrumental Activities of Daily comprises 8 items (ability to use the telephone, do the shopping, meal preparation, do the housework, do the laundry, use public transport, take responsibility for own medication and manage a budget.)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided